CLINICAL TRIAL: NCT05411198
Title: A Prospective, Multicenter Clinical Study to Evaluate the Safety and Effectiveness of Ab Externo Implantation of Glaucoma Gel Stent
Brief Title: Study to Assess Change in Disease Activity and Adverse Events of Ab Externo Approach for Glaucoma Gel Stent (XEN45) Implantation In Participants Aged 45 Years or Older With Open-Angle Glaucoma
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1924-703-007
Record Dates: First submitted 2022-06-06; First posted 2022-06-09 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Open-Angle Glaucoma
Keywords: Open-Angle Glaucoma; Glaucoma; OAG; XEN45; Glaucoma Gel Stent; XEN45 Glaucoma Treatment System
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- XEN45 (Glaucoma Gel Stent) (Experimental): Participants will receive XEN45 implanted using an ab externo approach on Day 1.
  Interventions: Device: XEN45 (Glaucoma Gel Stent)

INTERVENTIONS:
Device: XEN45 (Glaucoma Gel Stent) — Ab externo implant

SUMMARY:
Glaucoma is the second most common cause of blindness in the world, second only to cataracts. This study will assess how safe and effective a glaucoma gel stent is when implanted using the ab externo approach. Adverse events and intraocular pressure will be assessed.

XEN45 is an approved device for the treatment of glaucoma implanted using the ab interno approach (inside the eye). XEN45 implanted using the ab externo approach (outside the eye) is being studied in this study. Approximately 65 participants aged 45 years or older with open-angle glaucoma will be enrolled in this study at approximately 22 sites in the United States.

All participants will receive XEN45 implanted using the ab externo approach on Day 1 and will be followed for 12 months.

Participants will attend regular visits during the study at a hospital or clinic. The safety and effect of the gel stent on your glaucoma will be checked by medical assessments and eye examinations.

ELIGIBILITY:
Inclusion Criteria:

* Glaucoma in the study eye.

  1. Study eye diagnosed with open-angle glaucoma uncontrolled by medical therapy
  2. Study eye that meet at least one of the following criteria:

     * Failed one or more incisional intraocular glaucoma surgeries (e.g., glaucoma filtering surgery or tube shunt) (a minimum of approximately 15 subjects will be enrolled)
     * Failed one or more cilioablative procedures (e.g., cryotherapy, cyclodiode therapy)
     * Have neovascular glaucoma
     * Have any other condition (e.g., conjunctival scarring, uveitis) in which a conventional incisional glaucoma surgery like trabeculectomy would be more likely to fail than for a person with uncomplicated primary open-angle glaucoma (OAG).

     Note: To allow for a subgroup of participants who only have OAG uncontrolled by medical therapy (non-refractory glaucoma), a maximum of 10 participants who meet only criterion a (and not b) will be enrolled.

     Exclusion Criteria:
* A lack of healthy conjunctiva showing free mobility (free of scarring or evidence of prior surgery) in the target area.
* Excessive intraoperative bleeding, such that visualization in the study eye is impaired.
* Any anatomy or finding in the study eye that limits the investigator's ability to visualize the anterior chamber, angle, or target area of the conjunctiva.
* Other surgical complication that in the opinion of the investigator could impede proper placement of the Gel Stent.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2022-07-22 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Effectiveness of XEN45 | Month 12
  Effectiveness is defined as achieving 20% or more reduction of intraocular pressure (IOP) from baseline and on the same or fewer number of glaucoma medications than at baseline without secondary surgical intervention for IOP (SSII).

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (25):
- United States (23):
  - Vold Vision /ID# 245285, Fayetteville, Arkansas
  - UCLA Doheny Eye Center /ID# 227587, Pasadena, California
  - Ventura Ophthalmology /ID# 227585, Ventura, California
  - East Coast Institute for Research /ID# 255508, Jacksonville, Florida
  - Center for Sight - Sarasota /ID# 227577, Sarasota, Florida
  - New Vision Eye Center /ID# 261053, Vero Beach, Florida
  - Georgia Eye Partners /ID# 245203, Atlanta, Georgia
  - Stiles Eyecare Excellence /ID# 227576, Overland Park, Kansas
  - The Johns Hopkins Wilmer Eye Institute - Bethesda /ID# 245355, Bethesda, Maryland
  - Vance Thompson Vision /ID# 261125, Alexandria, Minnesota
  - Washington University-School of Medicine /ID# 245452, St Louis, Missouri
  - NYU Langone Medical Center /ID# 227583, New York, New York
  - Fichte Endl & Elmer Eyecare /ID# 245165, Niagara Falls, New York
  - Oklahoma Eye Surgeons /ID# 246840, Oklahoma City, Oklahoma
  - Ophthalmic Partners, PC /ID# 245367, Bala-Cynwyd, Pennsylvania
  - Kremer Eye Center - King of Prussia /ID# 245573, King of Prussia, Pennsylvania
  - Vance Thompson Vision /ID# 260892, Sioux Falls, South Dakota
  - Glaucoma Associates of Texas /ID# 227580, Dallas, Texas
  - University of Texas Southwestern Medical Center /ID# 246848, Dallas, Texas
  - El Paso Eye Surgeons, P.A. /ID# 227575, El Paso, Texas
  - Eye associates /ID# 227572, San Antonio, Texas
  - University of Utah /ID# 245324, Salt Lake City, Utah
  - Northern Virginia Ophthalmology Associates -Falls Church /ID# 246925, Falls Church, Virginia
- Australia (2):
  - Eye Surgery Associates /ID# 252207, East Melbourne, Victoria
  - Melbourne Eye Specialists /ID# 252353, Fitzroy, Victoria

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related info — https://www.rxabbvie.com/